CLINICAL TRIAL: NCT03843593
Title: Why Do Patients Agree To or Decline Adjuvant Immunotherapy and Are They Satisfied With Their Decision?
Brief Title: A Study To See Why Patients Agree To or Decline To Have Treatment After Surgery
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-012
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Cutaneous Melanoma
Keywords: Decline Adjuvant Immunotherapy; Agree To Adjuvant Immunotherapy; Nivolumab; Pembrolizumab; 19-012
MeSH Terms: conditions — Melanoma | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Melanoma patients: This is a pilot prospective study to identify the factors patients consider in deciding whether or not to undergo adjuvant therapy. Patients are eligible regardless of whether they decide to accept adjuvant therapy. If the researcher plans to treat the participant with pembrolizumab instead of nivolumab, it should be known that although the video discusses nivolumab, the risks and benefits are the same.
  Interventions: Behavioral: Demographics Questionnaire; Behavioral: Adjuvant Treatment Beliefs Scale10; Behavioral: Functional Assessment of Cancer Therapy - Melanoma (FACT-M)11; Behavioral: Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT-TS-G)13; Behavioral: Decisional Regret14; Behavioral: Clinician Preference for Treatment

INTERVENTIONS:
Behavioral: Demographics Questionnaire — A brief questionnaire will collect basic demographic information (i.e., age, gender, racial background, ethnicity, employment status, marital status) at time of enrollment.
Behavioral: Adjuvant Treatment Beliefs Scale10 — This brief PRO measure asks patients to indicate the likelihood, using a 5-point Likert type scale (1 [definitely not], 2 [probably not], 3 [maybe], 4 [probably], 5 [definitely]) of six positive (e.g., reduced risk of recurrence, greater chance of being cured) and five negative outcomes (e.g., side effects, health status) of adjuvant treatment.
Behavioral: Functional Assessment of Cancer Therapy - Melanoma (FACT-M)11 — FACT-M is a 51-item patient-self report measure for the assessment of quality of life (QOL) in patients with American Joint Committee on Cancer stages I through IV melanoma.
Behavioral: Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT-TS-G)13 — FACIT-TS-G is a brief, 8-item self-administered measure designed to assess general treatment satisfaction in patients.
Behavioral: Decisional Regret14 — This is a set of 5 questions examining level of regret for treatment decisions (in this case, decision to pursue adjuvant therapy), with answers scored on a 5-point Likert-type scale (i.e., 1 [Strongly Agree], 2 [Agree], 3 [Neither Agree Nor Disagree], 4 [Disagree], 5 [Strongly Disagree].
Behavioral: Clinician Preference for Treatment — This is a single item to be completed by Medical Oncologists that will indicate their preference as to whether they prefer that their patient accepts adjuvant therapy.

SUMMARY:
The purpose of this study is to find out what patients consider when deciding whether or not to receive adjuvant treatment, and how patients feel about their decision after one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IIIB, IIIC, IIID, or IV (AJCC, 8th edition) cutaneous melanoma rendered free of disease by surgical resection.
* Patients are being offered adjuvant nivolumab or pembrolizumab therapy
* Patient has not yet formally discussed their treatment options with their Medical Oncologist.
* Age 18 or older.
* Ability to speak and read English because we do not have the resources to translate materials into other languages.

Exclusion Criteria:

* Patient not currently free of disease.
* Candidate for adjuvant dabrafenib/trametinib therapy.
* Patients who have received prior checkpoint inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research participants will be identified by members of the Melanoma service, the patients" treatment team, or the PI.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
self-reported factors patients consider in deciding whether or not to undergo adjuvant therapy | 1 year
  Factors considered are gleaned from the Acceptance/Declination Survey

SECONDARY OUTCOMES:
self-reported quality of life | 1 year
  as captured by FACT-M, as well as treatment satisfaction. Functional Assessment of Cancer Therapy - Melanoma (FACT-M)11 - FACT-M is a 51- item patient-self report measure for the assessment of quality of life (QOL) in patients with American Joint Committee on Cancer stages I through IV melanoma.The FACT-M incorporates a recall period of 7-days and a five-point Likert-type scale (i.e., 0 = Not at all, 1 = A little bit, 2 = Somewhat, 3 = Quite a bit, 4 = Very much).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm